CLINICAL TRIAL: NCT05244993
Title: AK105 Plus Anlotinib Hydrochloride Combined With Albumin Paclitaxel as a First-line Therapy in Patients With Advanced Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Collaborators: Huludao central hospital (Unknown); Anshan Tumor Hospital (Other); Chaoyang Central Hospital (Other); Fukuang General Hospital of Liaoning health industry group (Unknown)
Responsible Party: Principal Investigator, Tao Sun, Director, Liaoning Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-BC-003
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK105+Anlotinib Hydrochloride+Albumin Paclitaxel (Experimental): AK105 200mg IV Day 1 Anlotinib Hydrochloride 12mg PO once daily on Days 1-14 Albumin paclitaxel 125mg/m2 IV Days 1, 8 Cycled every 21 days until disease progression, death or toxicity is intolerable (for subjects who can continue to tolerate the treatment, albumin paclitaxel lasts for at least 6 cycles)
  Interventions: Drug: AK105; Drug: Anlotinib hydrochloride; Drug: Albumin Paclitaxel

INTERVENTIONS:
Drug: AK105 — AK105: 100mg per bottle, 200mg IV Day 1, cycled every 21 days
  Other Names: Penpulimab
Drug: Anlotinib hydrochloride — Anlotinib Hydrochloride: 12mg per capsule, 12 mg PO once daily on Days 1-14, cycled every 21 days
Drug: Albumin Paclitaxel — Albumin paclitaxel: 100mg per bottle, 125mg/m2 IV Days 1, 8, cycled every 21 days

SUMMARY:
This trial used a multicentre, single-arm design in which patients were treated with AK105 plus Anlotinib Hydrochloride combined with albumin paclitaxel. Patients included in this trial were advanced breast cancer with hormone receptor negative and Her2 negative. The primary endpoint is ORR, and the secondary endpoint is DCR, PFS, OS and safety.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-75 years old.
* ECOG 0 or 1 point.
* Advanced triple-negative invasive breast cancer :

  1. The pathological classification is triple negative, specifically:

     1. ER negative: IHC<1%.
     2. PR negative: IHC<1%.
     3. HER2 negative: IHC-/+ or IHC++ but FISH/CISH is negative.
  2. Tumor staging: locally advanced or recurrent/metastatic breast cancer.
* If the last chemotherapy drug in the previous adjuvant/neoadjuvant treatment stage is paclitaxel, paclitaxel liposome, paclitaxel albumin or docetaxel, it will take ≥6 months from the end of treatment to enrollment.
* At least one objectively measurable lesion according to the RECIST 1.1 .
* The main organs are functioning well, and the blood test results within 14 days before enrollment should meet the following requirements:

  1. Routine blood test:

     1. Hemoglobin (HB) ≥90 g/L.
     2. Neutrophil count (ANC) ≥1.5×109/L.
     3. Platelet count (PLT) ≥100×109/L.
  2. Biochemical test:

     1. Total bilirubin≤1.5×ULN (upper limit of normal).
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; if there is liver metastasis, ALT and AST ≤ 5×ULN.
     3. Serum creatinine (Cr) ≤1.5 ULN or creatinine clearance ≥60mL/min.
* Must not be regnant.
* Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

* Pregnant, lactating or planning to become pregnant during the study period.
* Allergic to any of the drugs in the study.
* Previously received PD-1/PD-L1 antibody, CTLA-4 antibody, or anti-vascular targeted therapy.
* Central nervous system (CNS) metastases.
* Concomitant disease/medical history:

  1. Patients with any known or suspected autoimmune diseases.
  2. Hypertension.
  3. Peripheral neuropathy ≥ Grade 2.
  4. Persons with a history of unstable angina or arrhythmia.
  5. Active or uncontrolled serious infection .
  6. History of immunodeficiency.
  7. Active hepatitis B or C.
  8. interstitial lung disease or non-infectious pneumonia.
  9. Active tuberculosis.
  10. Urine protein is ≥++, and 24-hour urine protein quantitative is >1.0g.
  11. Suffered from other malignant tumors within 5 years before enrollment.
  12. Unreduced toxicity .
  13. Multiple factors that affect oral medications.
  14. Abnormal coagulation function.
  15. Major surgical treatment, open biopsy or traumatic injury within 4 weeks.
  16. Tumor has invaded the periphery of important blood vessels.
  17. Patients who have seizures.
  18. Bleeding constitution or medical history.
  19. Arterial/venous thrombotic events before enrollment or within 6 months.
  20. Live attenuated vaccine vaccination within 28 days before the study.
  21. Uncontrollable pleural, abdominal or pericardial effusion.
  22. Other uncontrollable systemic diseases.
* Other serious physical or mental diseases or laboratory abnormalities.
* Patients who the researcher thinks are not suitable for this research.
* Participated in clinical trials of other anti-tumor drugs within four weeks.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 10 months
  Overall response rate (ORR) is defined as the proportion of patients with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 10 months
  DCR: Disease Control Rate, defined as the proportion of patients with the best overall response of complete response (CR) , partial response (PR) or stable disease (SD) according to RECIST 1.1.
Progression Free Survival (PFS) | Up to approximately 10 months
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause.
Overall Survival (OS) | Up to approximately 18 months
  OS: Time from date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Doctor, Principal Investigator — Liaoning Cancer Hospital & Institute